CLINICAL TRIAL: NCT00987207
Title: Pharmacological Postconditioning During the Aortic Valvular Surgery
Acronym: PC Pharma CVA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007.490
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2011-11

CONDITIONS: Aortic Valvular Surgery
Keywords: Postconditioning; cyclosporine A; myocardial ischemia; cardiac surgery; aortic valvulopathy
MeSH Terms: conditions — Myocardial Ischemia | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- cyclosporine (Experimental): A single bolus of 2.5 mg/kg cyclosporine is administered before aortic cross-declamping
  Interventions: Drug: cyclosporine A
- Control (Other): No cyclosporine A is administered before aortic cross-declamping
  Interventions: Other: No injection

INTERVENTIONS:
Drug: cyclosporine A — a single bolus of 2.5 mg/kg, administered before aortic cross-declamping
  Arms: cyclosporine
Other: No injection — No cyclosporine A is administered before aortic cross-declamping.
  Arms: Control

SUMMARY:
Primary objective: To evaluate the efficacy of the cyclosporin A administration to induce a cardioprotection during the valvular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or females, scheduled for an aortic valvular surgery;
* 18 years of age or older.

Exclusion Criteria:

* Combined valvular and coronary surgery;
* Significant coronary artery stenosis (upper than 70%);
* Left ventricular dysfunction (ejection fraction < 40%);
* Emergency surgery and/or infectious endocarditis;
* Known cyclosporin hypersensitivity;
* History of known recent immunosuppression (< 6 months): cancer, lymphoma, positive serology for HIV, hepatitis;
* Renal insufficiency (creatininaemia > 150 µmol/l);
* Hepatic insufficiency (prothrombin time < 50%);
* Uncontrolled arterial hypertension defined by a systolic arterial pressure > 180 mm Hg;
* Women of child bearing potential, who are pregnant or not under efficient contraception;
* Patients treated with nicorandil, sulfonylurea or rosuvastatine;
* Patients under judicial control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The peak of the cardiac troponin I blood level measured during the first 72 hours of surgery follow-up. | 72 hours

SECONDARY OUTCOMES:
Area under curve of the cardiac troponin I release, BNP, length of mechanical ventilation, length of stay in ICU, SAPS, necessity of a catecholaminergic support to assure hemodynamic stability, SAE | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pascal CHIARI, MD, Principal Investigator — Hospices Civils de Lyon, France
Locations (1):
- Hôpital Louis Pradel, Lyon, France

REFERENCES:
- [Result] Chiari P, Angoulvant D, Mewton N, Desebbe O, Obadia JF, Robin J, Farhat F, Jegaden O, Bastien O, Lehot JJ, Ovize M. Cyclosporine protects the heart during aortic valve surgery. Anesthesiology. 2014 Aug;121(2):232-8. doi: 10.1097/ALN.0000000000000331. PMID 25050491